CLINICAL TRIAL: NCT05126511
Title: Effects of Cranial Electrotherapy Stimulation on Anxiety of Patients After COVID-19 - a Randomised Controlled Pilot Study
Brief Title: Effects of Cranial Electrotherapy Stimulation on Anxiety of Patients After COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Schön Klinik Berchtesgadener Land (Other)
Responsible Party: Principal Investigator, Prof. Dr. Andreas Rembert Koczulla, Head of Pneumological Department Affiliation: Schön Klinik Berchtesgadener Land, Schön Klinik Berchtesgadener Land
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AlphaStim
Record Dates: First submitted 2021-11-17; First posted 2021-11-19 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: POST-Covid 19; Anxiety
Keywords: Long-Covid/ Post-Covid; CES; fatigue; insomnia
MeSH Terms: conditions — Anxiety Disorders; Fatigue; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Post-Covid patients, anxious, functional device (Active Comparator): Applitation of 100µA CES for one hour per day to anxious patients
  Interventions: Device: Application of CES via ear clips
- Post-Covid patients, anxious, Sham (Placebo Comparator): Use of Sham CES for one hour per day by anxious patients
  Interventions: Device: Sham: No application of CES via ear clips
- Post-Covid patients, non anxious, functional device (Active Comparator): Application of 100µA CES for one hour per day to non anxious patients
  Interventions: Device: Application of CES via ear clips
- Post-Covid patients, non anxious, Sham (Placebo Comparator): Use of Sham CES for one hour per day by non anxious patients
  Interventions: Device: Sham: No application of CES via ear clips

INTERVENTIONS:
Device: Application of CES via ear clips — Use of 100µA CES for one hour per day over PR program
  Arms: Post-Covid patients, anxious, functional device; Post-Covid patients, non anxious, functional device
Device: Sham: No application of CES via ear clips — Use of Sham CES for one hour per day over PR programm
  Arms: Post-Covid patients, anxious, Sham; Post-Covid patients, non anxious, Sham

SUMMARY:
The aim of the study is to investigate the effect of cranial electrotherapy stimulation (CES), for one hour a day over 3 weeks pulmonary rehabilitation (PR) program on symptoms of anxiety in post-Covid patients.

DETAILED DESCRIPTION:
Many patients recovering from Covid-19 develop sequelae related to the disease. In addition to lung issues, symptoms of Post-Covid/Long-Covid Syndrome include fatigue, brain fog, amyosthenia, insomnia, anxiety and depression. These symptoms play a major role in post-Covid patients recovery.

CES (Cranial electrotherapy stimulation) is a non-invasive therapy using low intensity alternating current applied through electrodes attached to the ear lobe.

CES has been used to improve the condition of non covid patients suffering from depression, anxiety, fatigue and cognitive disabilities. This is thought to be due to a change in electric waves of the brain with an increase of alpha-waves and a decrease of beta- and delta-waves, as well as a change of concentration of neurotransmitters, e.g. beta-endorphin or serotonin.

Therefore, this study aims to investigate the effect of CES in addition to normal PR, compared to PR alone on symptoms (e.g. anxiety) in post-Covid patients.

Hypothesis: Three weeks of PR including daily use of CES for one hour will have a positive effect on symptoms of anxiety.

Trial: 40 patients post-Covid reffered to inpatient PR will be recruited and allocated to one of two different groups. Group1: Anxious participants, Group 2: Non anxious participants. Within groups particpants will be randomized to intervention or control/sham. Intervention group will be using a functional device, and the other using a non-functional, SHAM device.

Anxiety is evaluated using the Beck anxiety inventory on admission and at discharge from PR.

Questionnaires to evaluate fatigue, depression and insomnia are the Fatigue Assessment Scale, PHQ-9, PSQI).

A diary will be kept by each participant with a log of general health and mood over the PR program.

ELIGIBILITY:
Inclusion Criteria:

Group with anxiety:

* high Beck Anxiety Inventory Score
* ≥18 years
* post SARS-CoV-2 infection
* written consent

Group without anxiety:

* low Beck Anxiety Inventory Score
* ≥18 years
* post SARS-CoV-2 infection
* written consent

Exclusion Criteria:

* acitve implants (cardiac pacemaker,...)
* pregnancy, lactation period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-11-19 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Change of symptoms of anxiety during intervention | Day 1 and Day 21
  Comparison of the Beck Anxiety Inventory pre and post pulmonary rehabilitation

SECONDARY OUTCOMES:
Change in insomnia during intervention | Day 1 and Day 21
  Comparison of the PSQI questionnaire pre and post pulmonary rehabilitation
Change in fatigue during intervention | Day 1 and Day 21
  Comparison of the FAS questionnaire pre and post pulmonary rehabilitation
Change in depression during intervention | Day 1 and Day 21
  Comparison of the PHQ-9 questionnaire pre and post pulmonary rehabilitation
Change of general condition/ perceived well-being of the patient | Day 1 until Day 21
  Evaluation of the diary kept by the patient
Subjective effectiveness of device | Day 21
  Evaluation of the diary kept by the patient
Comfort while using the device | Day 21
  Evaluation of the diary kept by the patient

CONTACTS AND LOCATIONS:
Locations (1):
- Klinikum Berchtesgadener Land, Schön Kliniken, Schönau am Königssee, Bavaria, Germany